CLINICAL TRIAL: NCT05748600
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Efficacy, Safety, and Tolerability of Dexpramipexole Administered Orally for 24 Weeks in Participants With Eosinophilic Asthma
Brief Title: A Study to Assess the Effect of Dexpramipexole in Adolescents and Adults With Eosinophilic Asthma
Acronym: EXHALE-4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Areteia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR-DEX-22-03; 2022-003005-30 (EudraCT Number)
Record Dates: First submitted 2023-02-20; First posted 2023-02-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Eosinophilic Asthma; Asthma; Eosinophilic; Asthma Attack
Keywords: FEV1; Asthma; Dexpramipexole; EXHALE; EXHALE-4; Areteia; Uncontrolled Asthma; Asthma Attack; forced expiratory volume
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 150 mg BID (Experimental): Dexpramipexole 150 mg oral tablet taken twice a day
  Interventions: Drug: Dexpramipexole Dihydrochloride
- 75 mg BID (Experimental): Dexpramipexole 75 mg oral tablet taken twice a day
  Interventions: Drug: Dexpramipexole Dihydrochloride
- Placebo (Placebo Comparator): Placebo oral tablet taken twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexpramipexole Dihydrochloride — administration of dexpramipexole tablet
  Arms: 150 mg BID; 75 mg BID
Drug: Placebo — administration of placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate dexpramipexole as an add-on oral therapy in participants with inadequately controlled eosinophilic asthma to evaluate improvements in lung function, asthma control, and quality of life. In addition, the study will further evaluate the safety and tolerability of dexpramipexole in participants with eosinophilic asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form and assent form, as appropriate.
2. Male or female ≥12 years of age at Screening Visit 1. Sites in Poland will only include participants aged ≥18 years.

   Asthma-related criteria
3. Documented physician diagnosis of asthma for ≥12 months prior to Screening Visit 1.
4. Participants requiring at a minimum daily low dose inhaled corticosteroids (ICS; ≥100 μg/day fluticasone propionate dry powder formulation daily or clinically comparable, per GINA 2021), plus one or more additional daily maintenance asthma controller medications, eg, long-acting β2 agonist (LABA), leukotriene antagonist, theophylline, long-acting muscarinic antagonists, cromolyn/nedocromil. Note: In Poland, this will instead include participants requiring a minimum daily medium dose ICS (≥500 μg/day fluticasone propionate dry powder formulation daily or clinically comparable, per GINA 2021). Use of daily ICS must be for at least 12 weeks prior to Screening Visit 1 and the doses of all controller medications must be stable for at least 4 weeks prior to Screening Visit 1.
5. Pre-BD FEV1 ≥40% and <80% (<90% for participants 12 to 17 years of age) of predicted at Screening Visit 2.
6. Bronchodilator reversibility, at Screening Visit 2, as evidenced by ≥12% and ≥200 mL improvement in FEV1, 15 to 30 minutes following inhalation of 400 μg (four puffs) of albuterol/salbutamol (≥12% and ≥160 mL for ages 12 to 17).Participants who do not meet the bronchodilator reversibility inclusion criterion but have ≥10% and ≥160 mL reversibility, may repeat the reversibility spirometry assessment once during the Screening Period, at an unscheduled visit at least 7 days prior to baseline.
7. ACQ-6 ≥1.5 at Screening Visit 2.
8. Eosinophil count of ≥0.30x10⁹/L at Screening Visit 1. If the initial value is between 0.250x10⁹/L to 0.299x10⁹/L, then this may be repeated once at an unscheduled visit (prior to Screening Visit 2).

   General medical history
9. Negative urine pregnancy test for women of childbearing potential (WOCBP; after menarche) at the Screening and Baseline visits.
10. WOCBP must use either of the following methods of birth control, from Screening Visit 1 through the End of Study Visit:

    1. A highly effective form of birth control (confirmed by the investigator). Highly effective forms of birth control include: true sexual abstinence, a vasectomized sexual partner, Implanon, female sterilization by tubal occlusion, any effective intrauterine device (IUD), IUD/intrauterine system (IUS), Levonorgestrel Intrauterine system, or oral contraceptive.

       Or
    2. Two protocol acceptable methods of contraception in tandem.

       * Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months prior to the planned date of the Baseline Visit without an alternative medical cause. The following age specific requirements apply:
    3. Women <50 years old will be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone levels in the postmenopausal range.
    4. Women ≥50 years old will be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment. least 7 days prior to baseline.

Exclusion Criteria:

Asthma-related criteria

1. A participant who experiences a severe asthma exacerbation (defined as a deterioration of asthma that results in emergency treatment, hospitalization prior to the Screening Visit 1 up to and including the Baseline Visit.

   Participants who experience an asthma exacerbation during the Screening/Run-in Period may remain in screening and proceed with study visits 14 days after they have completed their course of oral steroids or returned to their pre-Screening visit maintenance dose of oral steroids and the investigator considers participant has returned to baseline status.
2. Current diagnosis of diseases which may confound interpretation of this study's findings such as allergic bronchopulmonary aspergillosis, eosinophilic granulomatosis with polyangiitis, eosinophilic gastrointestinal diseases, or hypereosinophilic syndrome, or lung diseases (eg, chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis).
3. Respiratory infection: Upper or lower respiratory tract, sinus, or middle ear infection within the 4 weeks before Screening Visit 1.

   Prohibited medications/procedures
4. Treatment with a biologic investigational drug in the last 5 months prior to Screening Visit 1. Treatment with non-biologic investigational drugs in the previous 30 days or five-half-lives prior to Screening Visit 1, whichever is longer. Treatment with GSK3511294 (long acting anti-interleukin-5) in the past 12 months.
5. Treatment with any of the following monoclonal antibody therapies within 120 days prior to Baseline: benralizumab, dupilumab, mepolizumab, reslizumab, omalizumab, tezepelumab, or tralokinumab.
6. Treatment with pramipexole (Mirapex®) within 30 days of Baseline.
7. Treatment with selected drugs known to have a substantial risk of neutropenia in the past 30 days prior to Screening Visit 1.
8. Bronchial thermoplasty procedure in the past 12 months prior to Screening Visit 1 or planned during the study period.

   General medical history
9. Weight <40 kg at Screening Visit 2.
10. Current smoking within 12 months prior to Screening Visit 1 or a smoking history of >10 packyears. Smoking includes tobacco, vaping, and/or marijuana use.
11. Known or suspected alcohol or drug abuse.
12. Uncontrolled severe hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg prior to the Baseline Visit despite antihypertensive therapy.
13. History of malignancy that required surgery (excluding local and wide-local excision), radiation therapy and/or systemic therapy during the 5 years prior to the Baseline Visit.
14. History of human immunodeficiency virus (HIV) infection or chronic infection with hepatitis B or C.
15. A helminth parasitic infection diagnosed within 24 weeks prior to Screening Visit 1, that has not been treated with or has failed to respond to standard of care therapy.
16. Medical or other condition likely to interfere with participant's ability to undergo study procedures, adhere to visit schedule, or comply with study requirements.
17. Known or suspected noncompliance with medication.
18. Unwillingness or inability to follow the procedures outlined in the protocol.

    Clinical safety labs
19. Absolute neutrophil count <2.000x10⁹/L at Screening Visit 1 or Screening Visit 2..
20. Renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 at Screening Visit 2 (using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula [Levey et al, 2009] for age ≥18 years at screening; using the Bedside Schwartz [Schwartz and Work, 2009] eGFR formula for age <18).
21. Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained elevations in alanine aminotransferase (ALT), aspartate aminotransferase (AST), >3x the upper limit of normal (ULN), or total bilirubin >2x ULN at Screening Visit 2 confirmed by a repeat abnormal measurement of the relevant value(s), at least 1 week apart.

    Cardiac safety
22. History of New York Heart Association class IV heart failure or last known left ventricular ejection fraction <25%.
23. History of major adverse cardiovascular event (MACE) within 3 months prior to the Baseline Visit.
24. History of cardiac arrhythmia within 3 months prior to the Baseline Visit that is not controlled by medication or via ablation.
25. History of long QT syndrome.
26. Corrected QT interval by Fridericia (QTcF) interval >450 ms for males and >470 ms for females at Screening Visit 2 or QTcF ≥480 ms for participants with bundle branch block.
27. Clinically important abnormalities in resting ECG that may interfere with the interpretation of QTcF interval changes at Screening Visit 2, including resting heart rate <45 beats per minute (bpm) or >100 bpm.

    Pregnancy/Lactation
28. Pregnant women or women breastfeeding.
29. Males who are unwilling to use an acceptable method of birth control during the entire study period (ie, condom with spermicide).

For this study, rescreening may only be permitted under specific circumstances and only after contact with a Sponsor Clinical representative.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in pre-BD FEV₁ from baseline | Day 1 (baseline, pre-dose), Weeks 20, 24
  Pre-bronchodilator forced expiratory volume (pre-BD) FEV₁, absolute change from baseline, averaged over Weeks 20 and 24.

SECONDARY OUTCOMES:
Change from baseline in Asthma Control Questionnaire-6 (ACQ-6) | Day 1 (baseline, pre-dose), Weeks 20, 24
  Change from baseline in Asthma Control Questionnaire-6 (ACQ-6) averaged over visits at Weeks 20 and 24.
Change in Standardized version of the Asthma Quality of Life Questionnaire for 12 years and older (AQLQ+12) from baseline to Week 24. | Day 1 (baseline, pre-dose) through Week 24
Change from baseline absolute eosinophil count (AEC) averaged across Weeks 20 and 24. | Day 1 (baseline, pre-dose) through Week 24
Change from baseline forced vital capacity (FVC) averaged over Weeks 20 and 24. | Day 1 (baseline, pre-dose), Weeks 20, 24
Change from baseline forced vital capacity (FVC) at Weeks 4, 8, 12, 16, 20, and 24. | Day 1 (baseline, pre-dose), Weeks 4, 8, 12, 16, 20, and 24
Change from baseline post-bronchodilator (post-BD) forced expiratory volume (FEV₁) at Week 24. | Day 1 (baseline, pre-dose) through Week 24
The EuroQol 5-dimensional questionnaire (EQ-5D-5L) change from baseline to Week 24 | Day 1 (baseline, pre-dose) through Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Mona Bafadhel, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (335):
- United States (146):
  - Research Site 40001-487, Chandler, Arizona
  - Research Site 40001-462, Peoria, Arizona
  - Research Site 40001-322, Surprise, Arizona
  - Research Site 40001-374, Bakersfield, California
  - Research Site 40001-227, Encinitas, California
  - Research Site 40001-349, Huntington Beach, California
  - Research Site 40001-485, Inglewood, California
  - Research Site 40001-440, La Palma, California
  - Research Site 40001-357, Lancaster, California
  - Research Site 40001-089, Los Angeles, California
  - Research Site 40001-362, Mission Viejo, California
  - Research Site 40001-449, Napa, California
  - Research Site 40001-062, Newport Beach, California
  - Research Site 40001-043, Newport Beach, California
  - Research Site 40001-380, Redding, California
  - Research Site 40001-434, San Diego, California
  - Research Site 40001-088, San Jose, California
  - Research Site 40001-359, Upland, California
  - Research Site 40001-003, West Covina, California
  - Research Site 40001-419, Westminster, California
  - Research Site 40001-425, Aurora, Colorado
  - Research Site 40001-353, Colorado Springs, Colorado
  - Research Site 40001-385, Wheat Ridge, Colorado
  - Research Site 40001-048, Aventura, Florida
  - Research Site 40001-005, Brandon, Florida
  - Research Site 40001-051, Brandon, Florida
  - Research Site 40001-029, Coral Gables, Florida
  - Research Site 40001-350, Gainesville, Florida
  - Research Site 40001-014, Greenacres City, Florida
  - Research Site 40001-054, Hialeah, Florida
  - Research Site 40001-067, Hialeah, Florida
  - Research Site 40001-020, Homestead, Florida
  - Research Site 40001-015, Kissimmee, Florida
  - Research Site 40001-002, Kissimmee, Florida
  - Research Site 40001-086, Loxahatchee Groves, Florida
  - Research Site 40001-318, Maitland, Florida
  - Research Site 40001-066, Miami, Florida
  - Research Site 40001-001, Miami, Florida
  - Research Site 40001-059, Miami, Florida
  - Research Site 40001-026, Miami, Florida
  - Research Site 40001-288, Miami, Florida
  - Research Site 40001-065, Miami, Florida
  - Research Site 40001-024, Miami, Florida
  - Research Site 40001-338, Miami Beach, Florida
  - Research Site 40001-348, Ocala, Florida
  - Research Site 40001-293, Orlando, Florida
  - Research Site 40001-429, Plantation, Florida
  - Research Site 40001-351, Sarasota, Florida
  - Research Site 40001-069, St. Petersburg, Florida
  - Research Site 40001-370, Tallahassee, Florida
  - Research Site 40001-004, Tampa, Florida
  - Research Site 40001-319, Viera, Florida
  - Research Site 40001-142, Adairsville, Georgia
  - Research Site 40001-075, Augusta, Georgia
  - Research Site 40001-018, Columbus, Georgia
  - Research Site 40001-452, Dunwoody, Georgia
  - Research Site 40001-483, East Point, Georgia
  - Research Site 40001-366, Lilburn, Georgia
  - Research Site 40001-423, Savannah, Georgia
  - Research Site 40001-090, Berwyn, Illinois
  - Research Site 40001-343, Chicago, Illinois
  - Research Site 40001-358, Normal, Illinois
  - Research Site 40001-135, River Forest, Illinois
  - Research Site 40001-403, Skokie, Illinois
  - Research Site 40001-036, Elwood, Indiana
  - Research Site 40001-347, Louisville, Kentucky
  - Research Site 40001-019, Owensboro, Kentucky
  - Research Site 40001-437, Alexandria, Louisiana
  - Research Site 40001-313, Marrero, Louisiana
  - Research Site 40001-352, Zachary, Louisiana
  - Research Site 40001-417, Annapolis, Maryland
  - Research Site 40001-466, Baltimore, Maryland
  - Research Site 40001-456, Takoma Park, Maryland
  - Research Site 40001-055, White Marsh, Maryland
  - Research Site 40001-468, Fall River, Massachusetts
  - Research Site 40001-427, Dearborn, Michigan
  - Research Site 40001-006, Flint, Michigan
  - Research Site 40001-148, Flint, Michigan
  - Research Site 40001-463, Rochester Hills, Michigan
  - Research Site 40001-442, Southfield, Michigan
  - Research Site 40001-372, Warren, Michigan
  - Research Site 40001-421, Mankato, Minnesota
  - Research Site 40001-083, Columbia, Missouri
  - Research Site 40001-074, Saint Charles, Missouri
  - Research Site 40001-046, St Louis, Missouri
  - Research Site 40001-409, Missoula, Montana
  - Research Site 40001-448, Lincoln, Nebraska
  - Research Site 40001-404, Omaha, Nebraska
  - Research Site 40001-473, Las Vegas, Nevada
  - Research Site 40001-387, Brick, New Jersey
  - Research Site 40001-363, Edison, New Jersey
  - Research Site 40001-457, Jersey City, New Jersey
  - Research Site 40001-355, Toms River, New Jersey
  - Research Site 40001-050, East Amherst, New York
  - Research Site 40001-412, Great Neck, New York
  - Research Site 40001-047, Hawthorne, New York
  - Research Site 40001-455, New York, New York
  - Research Site 40001-369, New York, New York
  - Research Site 40001-408, Charlotte, North Carolina
  - Research Site 40001-398, Charlotte, North Carolina
  - Research Site 40001-039, Gastonia, North Carolina
  - Research Site 40001-435, Greenville, North Carolina
  - Research Site 40001-111, Huntersville, North Carolina
  - Research Site 40001-382, Raleigh, North Carolina
  - Research Site 40001-439, Rocky Mount, North Carolina
  - Research Site 40001-283, Winston-Salem, North Carolina
  - Research Site 40001-034, Cincinnati, Ohio
  - Research Site 40001-013, Cincinnati, Ohio
  - Research Site 40001-010, Cincinnati, Ohio
  - Research Site 40001-413, Cleveland, Ohio
  - Research Site 40001-017, Dayton, Ohio
  - Research Site 40001-063, Toledo, Ohio
  - Research Site US-40001-038, Edmond, Oklahoma
  - Research Site 40001-386, Oklahoma City, Oklahoma
  - Research Site 40001-079, Oklahoma City, Oklahoma
  - Research Site 40001-027, Grants Pass, Oregon
  - Research Site 40001-337, Portland, Oregon
  - Research Site 40001-395, Hershey, Pennsylvania
  - Research Site 40001-327, Philadelphia, Pennsylvania
  - Research Site 40001-032, Columbia, South Carolina
  - Research Site 40001-025, Greenville, South Carolina
  - Research Site 40001-430, Rock Hill, South Carolina
  - Research Site 40001-073, Spartanburg, South Carolina
  - Research Site 40001-438, Dickson, Tennessee
  - Research Site 40001-414, Franklin, Tennessee
  - Research Site 40001-334, Allen, Texas
  - Research Site 40001-068, Amarillo, Texas
  - Research Site 40001-023, Dallas, Texas
  - Research Site 40001-028, Dallas, Texas
  - Research Site 40001-415, Dallas, Texas
  - Research Site 40001-304, DeSoto, Texas
  - Research Site 40001-418, Frisco, Texas
  - Research Site 40001-064, Houston, Texas
  - Research Site 40001-085, Houston, Texas
  - Research Site 40001-424, Kerrville, Texas
  - Research Site 40001-295, McKinney, Texas
  - Research Site 40001-304, Red Oak, Texas
  - Research Site 40001-377, San Antonio, Texas
  - Research Site 40001-335, Sugar Land, Texas
  - Research Site 40001-258, Murray, Utah
  - Research Site 40001-333, Pleasant View, Utah
  - Research Site 40001-340, Burke, Virginia
  - Research Site 40001-394, Williamsburg, Virginia
  - Research Site 40001-339, Greenfield, Wisconsin
  - Research Site 40001-433, La Crosse, Wisconsin
  - Research Site 40001-443, La Crosse, Wisconsin
- Argentina (16):
  - Research Site 40054-035, Buenos Aires
  - Research Site 40054-044, Buenos Aires
  - Research Site 40054-034, Buenos Aires
  - Research Site 40054-017, Buenos Aires
  - Research Site 40054-008, Buenos Aires
  - Research Site 40054-043, Buenos Aires
  - Research Site 40054-015, Caba
  - Research Site 40054-019, Mendoza
  - Research Site 40054-016, Mendoza
  - Research Site 40054-010, Mendoza
  - Research Site 40054-028, Mendoza
  - Research Site 40054-032, Mendoza
  - Research Site 40054-057, Mendoza
  - Research Site 40054-024, San Miguel de Tucumán
  - Research Site 40054-002, San Miguel de Tucumán
  - Research Site 40054-020, San Miguel de Tucumán
- Research Site 30043-013, Salzburg, Austria
- Brazil (13):
  - Research Site 40055-015, Belo Horizonte
  - Research Site 40055-007, Blumenau
  - Research Site 40055-011, Campo Largo
  - Research Site 40055-043, Curitiba
  - Research Site 40055-036, Curitiba
  - Research Site 40055-012, Porto Alegre
  - Research Site 40055-004, Porto Alegre
  - Research Site 40055-010, Porto Alegre
  - Research Site 40055-035, Rio de Janeiro
  - Research Site 40055-025, Salvador
  - Research Site 40055-005, Santo André
  - Research Site 40055-009, Santos
  - Research Site 40055-001, São Bernardo do Campo
- Canada (10):
  - Research Site 40011-004, Ajax, Ontario
  - Research Site 40011-016, Ajax, Ontario
  - Research Site 40011-010, Burlington, Ontario
  - Research Site 40011-014, Ottawa, Ontario
  - Research Site 40011-005, Windsor, Ontario
  - Research Site 40011-001, Windsor, Ontario
  - Research Site 40011-018, Montreal, Quebec
  - Research Site 40011-022, Québec, Quebec
  - Research Site 40011-020, Trois-Rivières, Quebec
  - Research Site 40011-011, Vancouver
- Israel (8):
  - Research Site 40972-010, Ashkelon
  - Research Site 40972-008, Beersheba
  - Research Site 40972-005, Haifa
  - Research Site 40972-004, Haifa
  - Research Site 40972-001, Jerusalem
  - Research Site 40972-009, Kfar Saba
  - Research Site 40972-002, Petah Tikva
  - Research Site 40972-011, Ramat Gan
- Research Site 30060-006, Kampung Kelantan, Malaysia
- Mexico (4):
  - Research Site 40052-026, Chihuahua City
  - Research Site 40052-007, Guadalajara
  - Research Site 40052-028, Mexico City
  - Research Site 40052-012, San Juan del Río
- Poland (23):
  - Research Site 40048-001, Będzin
  - Research Site 40048-018, Bialystok
  - Research Site 40048-032, Bialystok
  - Research Site 40048-023, Gdansk
  - Research Site 40048-006, Giżycko
  - Research Site 40048-021, Katowice
  - Research Site 40048-002, Katowice
  - Research Site 40048-027, Krakow
  - Research Site 40048-033, Krakow
  - Research Site 40048-008, Krakow
  - Research Site 40048-040, Krakow
  - Research Site 40048-015, Lodz
  - Research Site 40048-009, Lodz
  - Research Site 40048-005, Lodz
  - Research Site 40048-022, Lublin
  - Research Site 40048-024, Maków Podhalański
  - Research Site 40048-031, Ostrowiec Świętokrzyski
  - Research Site 40048-010, Piaseczno
  - Research Site 40048-016, Poznan
  - Research Site 40048-039, Rzeszów
  - Research Site 40048-014, Skierniewice
  - Research Site 40048-012, Trzebnica
  - Research Site 40048-019, Wroclaw
- Puerto Rico (7):
  - Research Site 40787-365, Guaynabo
  - Research Site 40787-390, Ponce
  - Research Site 40787-388, San Juan
  - Research Site 40787-383, San Juan
  - Research Site 40787-405, San Juan
  - Research Site 40787-360, San Juan
  - Research Site 40787-345, Vega Baja
- Romania (8):
  - Research Site 40040-004, Brasov, Brașov County
  - Research Site 40040-006, Cluj-Napoca, Cluj
  - Research Site 40040-002, Brasov
  - Research Site 40040-009, Cluj-Napoca
  - Research Site 40040-007, Cluj-Napoca
  - Research Site 40040-001, Constanța
  - Research Site 40040-010, Sângeorgiu de Mureş
  - Research Site 40040-003, Timișoara
- South Africa (19):
  - Research Site 40027-013, Benoni
  - Research Site 40027-025, Cape Town
  - Research Site 40027-009, Cape Town
  - Research Site 40027-011, Cape Town
  - Research Site 40027-021, Cape Town
  - Research Site 30090-020, Durban
  - Research Site 40027-007, Durban
  - Research Site 40027-026, Johannesburg
  - Research Site 40027-005, KwaZulu
  - Research Site 40027-008, KwaZulu
  - Research Site 40027-020, KwaZulu
  - Research Site 40027-023, KwaZulu
  - Research Site 40027-027, KwaZulu
  - Research Site 40027-010, KwaZulu
  - Research Site 40027-006, Mpumalanga
  - Research Site 40027-004, Pretoria
  - Research Site 40027-019, Pretoria
  - Research Site 40027-018, Vereeniging
  - Research Site 40027-017, Welkom
- South Korea (12):
  - Research Site 40082-003, Anyang-si
  - Research Site 30082-024, Bucheon-si
  - Research Site 40082-007, Busan
  - Research Site 40082-021, Gwangju
  - Research Site 40082-020, Incheon
  - Research Site 40082-006, Jeonju
  - Research Site 40082-019, Seoul
  - Research Site 40082-012, Seoul
  - Research Site 40082-008, Seoul
  - Research Site 40082-004, Seoul
  - Research Site 40082-011, Seoul
  - Research Site 40082-010, Suwon
- Taiwan (9):
  - Research Site 40886-001, Kaohsiung City
  - Research Site 40886-004, New Taipei City
  - Research Site 40886-006, New Taipei City
  - Research Site 40886-005, Taichung
  - Research Site 40886-007, Taichung
  - Research Site 40886-010, Taipei
  - Research Site 40886-008, Taipei
  - Research Site 40866-003, Taipei
  - Research Site 40886-009, Taipei
- Research Site 30066-004, Pathum Thani, Thailand
- Turkey (Türkiye) (18):
  - Research Site 40090-002, Adana
  - Research Site 40090-018, Ankara
  - Research Site 40090-021, Ankara
  - Research Site 40090-024, Ankara
  - Research Site 40090-003, Ankara
  - Research Site 40090-025, Ankara
  - Research Site 40090-008, Ankara
  - Research Site 40090-009, Ankara
  - Research Site 40090-017, Antalya
  - Research Site 40090-019, Bornova
  - Research Site 40090-020, Istanbul
  - Research Site 40090-026, Istanbul
  - Research Site 40090-011, Istanbul
  - Research Site 40090-012, Konak
  - Research Site 40090-016, Merkez
  - Research Site 40090-013, Mersin
  - Research Site 40090-024, Pendik
  - Research Site 40090-022, Tekirdağ
- Ukraine (21):
  - Research Site 40380-002, Chernivtsi
  - Research Site 40380-021, Chernivtsi
  - Research Site 40380-009, Ivano-Frankivsk
  - Research Site 40380-004, Ivano-Frankivsk
  - Research Site 40380-017, Ivano-Frankivsk
  - Research Site 40380-014, Ivano-Frankivsk
  - Research Site 40380-019, Kyiv
  - Research Site 40380-018, Kyiv
  - Research Site 40380-007, Kyiv
  - Research Site 40380-010, Kyiv
  - Research Site 40380-012, Kyiv
  - Research Site 40380-015, Kyiv
  - Research Site 40380-011, Kyiv
  - Research Site 40380-013, Kyiv
  - Research Site 40380-016, Lutsk
  - Research Site 40380-001, Ternopil
  - Research Site 40380-003, Vinnytsia
  - Research Site 40380-020, Vinnytsia
  - Research Site 40380-008, Vinnytsia
  - Research Site 40380-022, Vinnytsia
  - Research Site 40380-005, Zhytomyr
- United Kingdom (18):
  - Research Site 40044-018, Bellshill
  - Research Site 40044-021, Birmingham
  - Research Site 40044-077, Bollington
  - Research Site 40044-017, Chorley
  - Research Site 40044-022, Enfield
  - Research Site 40044-019, Liverpool
  - Research Site 40044-084, London
  - Research Site 40044-001, Manchester
  - Research Site 40044-020, Manchester
  - Research Site 40044-013, Manchester
  - Research Site 40044-009, Manchester
  - Research Site 40044-036, Manchester
  - Research Site 40044-006, Manchester
  - Research Site 40044-024, Preston
  - Research Site 40044-026, Rochdale
  - Research Site 40044-008, Salford
  - Research Site 40044-034, Stockport
  - Research Site 40044-078, Wythenshawe

IPD SHARING:
Plan to Share IPD: No